CLINICAL TRIAL: NCT00249873
Title: A Parallel Randomized Controlled Evaluation of Clopidogrel Plus Aspirin, With Factorial Evaluation of Irbesartan, for the Prevention of Vascular Events, in Patients With Atrial Fibrillation
Brief Title: Atrial Fibrillation Clopidogrel Trial With Irbesartan for Prevention of Vascular Events (ACTIVE A)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC4912 A
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Results first posted 2010-03-26 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Atrial Fibrillation; Vascular Risk
Keywords: Atrial fibrillation; Anticoagulant therapy; Thromboembolic prevention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel + ASA (Experimental): Clopidogrel 75 mg once daily (od) plus acetylsalicyclic acid (ASA) 75 to 100 mg od recommended (dose at the investigators' discretion)
  Interventions: Drug: clopidogrel (SR25990C)
- Placebo + ASA (Placebo Comparator): Matching placebo of clopidogrel 75 mg od plus acetylsalicyclic acid (ASA) 75 to 100 mg od recommended (dose at the investigators' discretion)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clopidogrel (SR25990C) — oral administration (tablets)
  Other Names: Plavix®
  Arms: Clopidogrel + ASA
Drug: placebo — oral administration (tablets)
  Arms: Placebo + ASA

SUMMARY:
The purpose of this study is to determine if the combination of clopidogrel 75mg once daily (od) plus aspirin 100mg daily (recommended dose) is better than aspirin alone (100mg daily recommended dose) for preventing vascular events such as stroke and heart attack during approximately three years of follow-up in patients with atrial fibrillation associated with at least one major risk factor of vascular event such as elderly, blood pressure increase, history of stroke or transient ischemic attack or left ventricular dysfunction etc. The study will also accept patients with atrial fibrillation and unwilling to take oral anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for ACTIVE A patients must have in same time the three following conditions :

* Evidence of atrial fibrillation either on one current Electrocardiogram (ECG) or two ECGs recorded at two weeks a part during 6 months prior to study enrollment.
* Evidence of high risk of vascular events : at least one of the following risk criteria must be present :

  * are 75 years greater;
  * on treatment for systemic hypertension;
  * prior stroke, Transient Ischemic Attack (TIA) or non-Central Nervous System (non-CNS) systemic embolus;
  * left ventricular dysfunction with left ventricular ejection fraction (EF) estimated by echocardiogram or angiogram (radionuclide or contrast) to be < 45%;
  * peripheral vascular disease (previous peripheral artery revascularization, limb and foot amputation, or the combination of current intermittent claudication and ankle arm systolic blood pressure ratio < 0.9);
  * age 55 to 74 years and either; f1) diabetes mellitus requiring drug therapy, or f2) documented previous myocardial infarction or documented coronary artery disease.
* To have either a contraindication to use an oral anticoagulant treatment or they are unwilling to take an oral anticoagulant treatment.

Exclusion Criteria:

Patients will be excluded from ACTIVE if any of the following are present :

* requirement for clopidogrel (such as recent coronary stent procedure)
* requirement for oral anticoagulant (such as prosthetic mechanical heart valve);
* prior intolerance to ASA or clopidogrel;
* documented peptic ulcer disease within the previous 6 months;
* prior intracerebral hemorrhage;
* significant thrombocytopenia; (platelet count < 50 x 10(9)/L)
* psychosocial reason making study participation impractical;
* geographic reason making study participation impractical;
* ongoing alcohol abuse;
* mitral stenosis,
* pregnant or nursing woman or woman of child bearing potential and not on effective birth control for at least one month prior to start of study or not willing to continue on birth control for duration of study; (severe comorbid condition such that the patient is not expected to survive 6 months;
* patient currently receiving an investigational pharmacologic agent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7554 (Actual)
Dates: Start 2003-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe YUSUF, Prof., Study Chair — Hamilton Health Sciences Corporation
Locations (30):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis, Vienna, Austria
- Sanofi-aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] ACTIVE Investigators; Connolly SJ, Pogue J, Hart RG, Hohnloser SH, Pfeffer M, Chrolavicius S, Yusuf S. Effect of clopidogrel added to aspirin in patients with atrial fibrillation. N Engl J Med. 2009 May 14;360(20):2066-78. doi: 10.1056/NEJMoa0901301. Epub 2009 Mar 31. PMID 19336502
- [Derived] Pare G, Mehta SR, Yusuf S, Anand SS, Connolly SJ, Hirsh J, Simonsen K, Bhatt DL, Fox KA, Eikelboom JW. Effects of CYP2C19 genotype on outcomes of clopidogrel treatment. N Engl J Med. 2010 Oct 28;363(18):1704-14. doi: 10.1056/NEJMoa1008410. Epub 2010 Aug 29. PMID 20979470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from June 2003 until May 2006. The study was conducted at 580 centers in 33 countries. The planned final follow-up visit date ensuring a median follow-up of three years was November 2008. The follow-up of the study was actually completed on March 2009 corresponding to an actual median follow-up of 3.5 years.
Groups:
- Placebo + ASA: Matching placebo of clopidogrel 75 mg od plus ASA 75 to 100 mg od recommended (dose at the investigators' discretion)
Period: Overall Study
Arm/Group | Clopidogrel + ASA | Placebo + ASA
Started | 3772 (randomized patients: patients remained in the study whether treated or not until planned study end) | 3782 (randomized patients: patients remained in the study whether treated or not until planned study end)
Completed | 2442 (started and completed study drug) | 2528 (started and completed study drug)
Not Completed | 1330 | 1254
Not completed — Not treated | 7 | 8
Not completed — Significant thrombocytopenia | 9 | 8
Not completed — Severe allergic reaction | 8 | 1
Not completed — Serious haemorrhagic Adverse Event | 74 | 30
Not completed — Other Serious Adverse Event | 86 | 97
Not completed — Qualifying condition not present | 20 | 23
Not completed — Contraindication to oral anticoagulant | 4 | 8
Not completed — Withdrawal by Subject | 504 | 466
Not completed — Lost to Follow-up | 4 | 7
Not completed — Minor bleeding | 99 | 37
Not completed — Non-compliance | 41 | 46
Not completed — Other non serious Adverse Event | 112 | 108
Not completed — Other contraindicated medication | 1 | 0
Not completed — Patient not wish to continue after May08 | 3 | 4
Not completed — Physician withdrew consent | 59 | 60
Not completed — Open label clopidogrel required | 31 | 42
Not completed — Angiotensin II receptor blocker required | 1 | 0
Not completed — Oral anticoagulant required | 159 | 157
Not completed — Study drug intolerance | 5 | 0
Not completed — Surgery/ procedure | 9 | 9
Not completed — Event related to cardiac condition | 12 | 21
Not completed — Thromboembolic/outcome event | 82 | 122

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel + ASA | Placebo + ASA | Total
Number analyzed (Participants) | 3772 | 3782 | 7554
Age, Customized [Number; unit: participants]
  18 to <65 years | 931 | 935 | 1866
  65 to <75 years | 1291 | 1258 | 2549
  >= 75 years | 1550 | 1589 | 3139
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (10.2) | 71.1 (10.2) | 71.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1560 | 1597 | 3157
  Male | 2212 | 2185 | 4397
CHADS2 Score [Number; unit: participants] — CHADS2 score is the Congestive heart failure, High blood pressure, Age, Diabetes, Stroke 2 score. It is a validated clinical prediction rule for determining the risk of stroke. It assigns points (0-6) depending on the presence or absence of co-morbidities such as history of Congestive heart failure, hypertension, Age, history of Diabetes, previous Stroke. A high score means higher risk of stroke.
  participants
    0 | 105 | 101 | 206
    1 | 1360 | 1338 | 2698
    2 | 1263 | 1315 | 2578
    >2 | 1040 | 1028 | 2068
    Missing | 4 | 0 | 4
Sitting Systolic Blood Pressure [Number; unit: participants]
  <120 mmHg | 603 | 620 | 1223
  >=120 mmHg | 3166 | 3159 | 6325
  Missing | 3 | 3 | 6
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 28.370 (5.575) | 28.459 (6.022) | 28.415 (5.803)

OUTCOME MEASURES:

1. Primary Outcome: First Occurence of Any Component of the Composite of Stroke, Non-Central Nervous System (Non-CNS) Systemic Embolism, Myocardial Infarction or Vascular Death as Per Adjudication
Description: The primary event is the first occurence of any adjudicated component of the following cluster over the duration of follow-up :
  * stroke (nonfatal or fatal)
  * myocardial infarction (nonfatal or fatal)
  * non-CNS systemic embolism
  * vascular death
  The primary efficacy analysis is performed on the time from randomization to this primary event. Numbers of patients with the composite event over the duration of the follow-up are presented by arm group.
Time Frame: expected median follow-up of approximately 3 years
Population: The intent-to-treat (ITT) population was used for all analyses. This consisted of all randomized patients irrespective of whether or not the patient actually received study drug or the patient's compliance with the study protocol. All patients were included in the treatment group to which they were originally allocated.
Measure: Number; unit: participants
Arm/Group | Clopidogrel + ASA | Placebo + ASA
Number analyzed (Participants) | 3772 | 3782
participants
  All components | 832 | 924
  - Myocardial Infarction (fatal or not) | 84 | 105
  - Stroke (fatal or not) | 285 | 391
  - Non-CNS systemic embolism | 50 | 48
  - Vascular death | 413 | 380
Statistical Analysis 1: Comparison: Clopidogrel + ASA vs Placebo + ASA; Test type: Superiority or Other; p = 0.0133, Log Rank — Cumulative incidence functions in each treatment group were calculated using non-parametric Kaplan-Meier estimates. Median time-to-event was not reached in any group. The primary comparison was performed at the 5% level using a 2-sided Log rank test; Hazard Ratio (HR) = 0.89, 95% CI [0.81 to 0.98] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of any component of the primary event for the clopidogrel group compared with the Placebo group

2. Secondary Outcome: Occurrence of Stroke
Description: The event is the occurence of stroke (nonfatal or fatal, ischemic, hemorrhagic or of uncertain type) after validation of the Event Adjudication Committee . The analysis is performed on the time from randomization to the occurrence of this event. Numbers of patients with the event over the duration of the follow-up are presented by arm group.
Time Frame: expected median follow-up of approximately 3 years
Population: The intent-to-treat (ITT) population was used for this analysis.
Measure: Number; unit: participants
Arm/Group | Clopidogrel + ASA | Placebo + ASA
Number analyzed (Participants) | 3772 | 3782
participants | 296 | 408
Statistical Analysis 1: Comparison: Clopidogrel + ASA vs Placebo + ASA; Test type: Superiority or Other; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI [0.62 to 0.83] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of stroke for the clopidogrel group compared with the Placebo group

3. Secondary Outcome: Death From Any Cause (Cardiovascular and Noncardiovascular)
Description: The considered event is death from any cause. The analysis is performed on the time from randomization to this event. Numbers of patients with the event over the duration of the follow-up are presented by arm group.
Time Frame: expected median follow-up of approximately 3 years
Population: The intent-to-treat (ITT) population was used for the analysis.
Measure: Number; unit: participants
Arm/Group | Clopidogrel + ASA | Placebo + ASA
Number analyzed (Participants) | 3772 | 3782
participants | 825 | 841
Statistical Analysis 1: Comparison: Clopidogrel + ASA vs Placebo + ASA; Test type: Superiority or Other; p = 0.696, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI [0.89 to 1.08] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of death from any cause for the clopidogrel group compared with the Placebo group

4. Secondary Outcome: Adjudicated Major Bleedings
Description: The number of participants with at least one major bleeding, validated by the Event Adjudication Committee are counted over the duration of the follow-up (including after permanent discontinuation of the study drug).
Time Frame: expected median follow-up of approximately 3 years
Population: The intent-to-treat (ITT) population was used for the analysis.
Measure: Number; unit: participants
Arm/Group | Clopidogrel + ASA | Placebo + ASA
Number analyzed (Participants) | 3772 | 3782
participants | 251 | 162
Statistical Analysis 1: Comparison: Clopidogrel + ASA vs Placebo + ASA; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: From randomization through 28 days after the end of study drug treatment or the final follow-up visit. In both treatment groups, median duration of exposure was approximately 36 months, with a maximum of 62 months.
Description: The intent to treat population was also used for safety analyses.
Arm/Group | Clopidogrel + ASA | Placebo + ASA
Serious Adverse Events (participants affected / at risk) | 1154/3772 | 1069/3782
Other Adverse Events (participants affected / at risk) | 2542/3772 | 2502/3782
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clopidogrel + ASA (N=3772) | Placebo + ASA (N=3782)
Anaemia (Blood and lymphatic system disorders) | 18 | 19
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 2
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 1
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 1
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 2 | 0
Hydrocele (Congenital, familial and genetic disorders) | 2 | 1
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 4
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 7
Vertigo positional (Ear and labyrinth disorders) | 2 | 2
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 0 | 1
Ectopic hyperthyroidism (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 3 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 9
Hypothyroidism (Endocrine disorders) | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 0 | 2
Angle closure glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 20 | 18
Corneal degeneration (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 2
Eyelid oedema (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 2 | 1
Maculopathy (Eye disorders) | 1 | 0
Pupils unequal (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 2
Retinal degeneration (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 3
Retinal haemorrhage (Eye disorders) | 1 | 1
Retinal vein thrombosis (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Abdominal strangulated hernia (Gastrointestinal disorders) | 3 | 0
Acute abdomen (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 3
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Colonic polyp (Gastrointestinal disorders) | 4 | 6
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 11 | 10
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 3 | 1
Diverticulum (Gastrointestinal disorders) | 4 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 5 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 6 | 7
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 2 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 3 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gallstone ileus (Gastrointestinal disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 8 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 21 | 6
Gastritis (Gastrointestinal disorders) | 8 | 7
Gastritis erosive (Gastrointestinal disorders) | 2 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 9 | 3
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 26 | 9
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 1
Gastrooesophagitis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 3 | 3
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 6 | 4
Inguinal hernia (Gastrointestinal disorders) | 18 | 17
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 1
Intestinal dilatation (Gastrointestinal disorders) | 0 | 1
Intestinal functional disorder (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 7 | 5
Intestinal perforation (Gastrointestinal disorders) | 4 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Intestinal strangulation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 3
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Mesenteric occlusion (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 8
Pancreatitis acute (Gastrointestinal disorders) | 1 | 4
Pancreatitis chronic (Gastrointestinal disorders) | 2 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 3
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 5 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 4 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 10 | 1
Rectal polyp (Gastrointestinal disorders) | 2 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 2
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 6 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 28 | 7
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 4
Asthenia (General disorders) | 2 | 3
Chest pain (General disorders) | 7 | 8
Cyst (General disorders) | 1 | 0
Death (General disorders) | 1 | 2
Dysplasia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Gait disturbance (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 7 | 4
Generalised oedema (General disorders) | 2 | 0
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 2
Multi-organ failure (General disorders) | 8 | 8
Non-cardiac chest pain (General disorders) | 3 | 8
Oedema peripheral (General disorders) | 2 | 0
Pelvic mass (General disorders) | 1 | 0
Perforated ulcer (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Puncture site haemorrhage (General disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 4
Submandibular mass (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 2
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 2
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 16 | 12
Cholecystitis acute (Hepatobiliary disorders) | 5 | 9
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 16 | 18
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 2
Hepatic congestion (Hepatobiliary disorders) | 0 | 3
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 2 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 2
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 2
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 2 | 0
Abscess neck (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
American trypanosomiasis (Infections and infestations) | 0 | 1
Anogenital warts (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 7 | 3
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 3 | 3
Bacterial infection (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0
Bronchiectasis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 20 | 13
Bronchitis viral (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 10 | 15
Cellulitis (Infections and infestations) | 9 | 7
Central line infection (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 2
Clostridial infection (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Corneal abscess (Infections and infestations) | 1 | 0
Cryptosporidiosis infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 2 | 0
Dengue fever (Infections and infestations) | 0 | 1
Dermo-hypodermitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 11 | 7
Emphysematous cholecystitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 5 | 10
Escherichia infection (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 2
Gangrene (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 13 | 10
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 2
Hepatitis e (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 2
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 3 | 4
Intervertebral discitis (Infections and infestations) | 1 | 0
Keratitis fungal (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 7 | 10
Localised infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 5 | 7
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 5 | 4
Meningitis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 2
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 3
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 2
Perirectal abscess (Infections and infestations) | 1 | 0
Peritoneal infection (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumococcal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 139 | 128
Pneumonia klebsiella (Infections and infestations) | 2 | 1
Pneumonia primary atypical (Infections and infestations) | 2 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 2
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Portal pyaemia (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 2 | 2
Post procedural sepsis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 3 | 2
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 5 | 10
Pyelonephritis acute (Infections and infestations) | 1 | 2
Renal abscess (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 8 | 6
Sepsis (Infections and infestations) | 27 | 19
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 6 | 10
Sinusitis (Infections and infestations) | 1 | 2
Skin bacterial infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Staphylococcal toxaemia (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tetanus (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Urethritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 23 | 28
Urosepsis (Infections and infestations) | 7 | 7
Viral infection (Infections and infestations) | 3 | 3
Viral pericarditis (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 4 | 4
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 4
Asbestosis (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 6 | 4
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 7
Ear injury (Injury, poisoning and procedural complications) | 0 | 1
Epiphyseal fracture (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 3
Fall (Injury, poisoning and procedural complications) | 24 | 19
Femoral neck fracture (Injury, poisoning and procedural complications) | 9 | 6
Femur fracture (Injury, poisoning and procedural complications) | 15 | 19
Foot fracture (Injury, poisoning and procedural complications) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 2 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 2 | 0
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 7 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 12 | 18
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 6 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 3
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 2 | 0
Open fracture (Injury, poisoning and procedural complications) | 1 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 3 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 2
Pharyngeal injury (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 10 | 10
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 9 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 4 | 6
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 14 | 3
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 2
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 9 | 8
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 4 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 3 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 7 | 4
Wound (Injury, poisoning and procedural complications) | 2 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 1
Aspiration bronchial (Investigations) | 0 | 1
Carbohydrate tolerance decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 3 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 19 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 4 | 3
Haemosiderosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 9
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 2
Starvation (Metabolism and nutrition disorders) | 1 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 9
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 28 | 36
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Senile osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 7
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 13
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 11
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cystosarcoma phyllodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 11
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritoneal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 16
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 4 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral disorder (Nervous system disorders) | 2 | 0
Cerebral haematoma (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cervical root pain (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 3 | 0
Convulsion (Nervous system disorders) | 3 | 4
Dementia (Nervous system disorders) | 4 | 3
Dementia Alzheimer's type (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 5 | 8
Dizziness postural (Nervous system disorders) | 1 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 5 | 4
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 1
Guillain-barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 3
Haemorrhagic stroke (Nervous system disorders) | 17 | 10
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 2 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 2
Intracranial haematoma (Nervous system disorders) | 0 | 1
Ivth nerve paralysis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0
Mononeuropathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
Parkinson's disease (Nervous system disorders) | 1 | 3
Polyneuropathy (Nervous system disorders) | 1 | 4
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 4
Radicular syndrome (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 2 | 2
Simple partial seizures (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 12 | 9
Syncope vasovagal (Nervous system disorders) | 1 | 4
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 1
Vascular encephalopathy (Nervous system disorders) | 4 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Bipolar i disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 6 | 5
Delirium (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0
Delusional disorder, persecutory type (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 11 | 5
Hallucination (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 2 | 1
Mental disorder (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1
Neurosis (Psychiatric disorders) | 0 | 1
Panic disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2
Schizophrenia (Psychiatric disorders) | 1 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder stenosis (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 2 | 2
Calculus urinary (Renal and urinary disorders) | 1 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 2 | 0
Cystitis ulcerative (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Enuresis (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 10 | 4
Haemorrhage urinary tract (Renal and urinary disorders) | 4 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Nephropathy (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 4 | 1
Renal cyst (Renal and urinary disorders) | 2 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 16 | 14
Renal failure acute (Renal and urinary disorders) | 22 | 23
Renal failure chronic (Renal and urinary disorders) | 3 | 5
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 3 | 4
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urethral fistula (Renal and urinary disorders) | 2 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 4 | 6
Urinary bladder haemorrhage (Renal and urinary disorders) | 2 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 11 | 2
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 12 | 13
Breast mass (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Colpocele (Reproductive system and breast disorders) | 0 | 1
Endometrial atrophy (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 2
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1
Prostatic disorder (Reproductive system and breast disorders) | 0 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 2
Prostatitis (Reproductive system and breast disorders) | 4 | 3
Prostatomegaly (Reproductive system and breast disorders) | 0 | 3
Rectocele (Reproductive system and breast disorders) | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 2 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Vaginal cyst (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 28 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Bedridden (Social circumstances) | 1 | 0
Disability (Social circumstances) | 0 | 1
Elderly (Social circumstances) | 1 | 0
Joint prosthesis user (Social circumstances) | 2 | 0
Social problem (Social circumstances) | 0 | 1
Social stay hospitalisation (Social circumstances) | 0 | 1
Circumcision (Surgical and medical procedures) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 1
Intestinal stoma (Surgical and medical procedures) | 0 | 1
Intraocular lens implant (Surgical and medical procedures) | 0 | 1
Obesity surgery (Surgical and medical procedures) | 1 | 0
Wound drainage (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 1 | 1
Angiodysplasia (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 6
Aortic aneurysm rupture (Vascular disorders) | 1 | 2
Aortic dissection (Vascular disorders) | 1 | 1
Aortic rupture (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 2
Cardiovascular insufficiency (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 3
Haemorrhage (Vascular disorders) | 6 | 3
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 5 | 3
Orthostatic hypotension (Vascular disorders) | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 1
Thrombosis (Vascular disorders) | 1 | 0
Varicose ulceration (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 2
Venous insufficiency (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clopidogrel + ASA (N=3772) | Placebo + ASA (N=3782)
Any Infections and infestations (Infections and infestations) | 994 | 961
Any Gastrointestinal disorders (Gastrointestinal disorders) | 806 | 763
Any Nervous system disorders (Nervous system disorders) | 661 | 682
Dizziness (Nervous system disorders) | 300 | 312
Any General disorders and administration site conditions (General disorders) | 582 | 541
Any Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 538 | 510
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 231 | 215
Any Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 532 | 623
Any Vascular disorders (Vascular disorders) | 440 | 414
Any Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 433 | 353
Any Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 337 | 289
Any Cardiac disorders (Cardiac disorders) | 301 | 314
Any Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 239 | 257
Any Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 220 | 208
Any Eye disorders (Eye disorders) | 190 | 198
Any Investigations (Investigations) | 185 | 201
Any Renal and urinary disorders (Renal and urinary disorders) | 184 | 196

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the study will be made jointly in the name of all wholehearted collaborators. Other papers will be authored based on the contributions of the individuals to the overall study. Substudies with scientific merit which have received prior approval from the Steering Committee (SC) may be published in the names of the contributing investigators. A copy of all manuscripts will be provided to the sponsors for their review. The final decision to publish articles will be made by the SC.